CLINICAL TRIAL: NCT06597994
Title: Therapy Optimisation Study of Adaptive Pudendal Neuromodulation in Women With Urinary Incontinence Implanted With the Amber UI System.
Brief Title: Augmenting Urinary Reflex Activity: Study 3
Acronym: AURA-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amber Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS-01388
Record Dates: First submitted 2024-08-09; First posted 2024-09-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amber UI Therapy (Experimental): Participants will receive optimised recharge accessories and device firmware upgrades
  Interventions: Device: Amber UI system

INTERVENTIONS:
Device: Amber UI system — Upgrade of Amber UI system recharge accessories and system firmware

SUMMARY:
AURA-3 study (Augmenting Urinary Reflex Activity Study 3) is a single arm, short-duration (8 month) cohort follow up study of preceding interventional medical device study, AURA-2.

ELIGIBILITY:
Inclusion Criteria:

* Participant has exited the AURA-2 clinical investigation.
* Participant has an implanted Amber UI system.
* Consents to participation.

Exclusion Criteria:

* Participant has withdrawn from AURA-2 clinical investigation.
* Participant is pregnant.
* A past or current condition that in the opinion of the PI contraindicates enrolment (PI discretion).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in absolute recharge performance | 48 hours; 2 weeks; 2 months; 2 months + 1 week; 4 months; 8 months
  Change in perceived recharge usability before and after receiving new recharge accessories and training.
Change in relative recharge performance | 48 hours; 2 weeks; 2 months; 2 months + 1 week; 4 months; 8 months
  Relative (percentage) change in frequency and duration of recharging sessions after receiving new recharge accessories and training compared to baseline.

SECONDARY OUTCOMES:
Change in recharge usability | 48 hours; 2 weeks; 2 months; 2 months + 1 week; 4 months; 8 months
  % of time the device is fully operational and available for use after receiving new recharge accessories and training compared to baseline
Fully adaptive mode usability | 48 hours; 2 months; 8 months
  Change in frequency, severity and impact on quality of life of urinary incontinence episodes as assessed by Short Form version of the International Consultation on Incontinence urinary questionnaire (ICIQ-UI SF) after receiving fully adaptive firmware update and training compared to baseline. The ICIQ-UI SF is a 4 item simple questionnaire with minimum value of 0 and maximum value of 21 with higher scores indicating higher severity of UI symptoms and their impact on health-related quality of life.
Fully adaptive mode specificity | 48 hours; 2 months; 8 months
  Change in quality of life in relation to change in obstructive symptoms, irritative symptoms and stress symptoms as assessed by the Long Form version of the Urogenital Distress Inventory (UDI-LF) after receiving fully adaptive firmware update and training compared to baseline. The UDI-LF consists of 19 questions and total scores are converted to a score range of 0-300, with higher scores representing greater symptom distress.
Adverse Device Events | 48 hours; 2 weeks; 2 months; 2 months + 1 week; 4 months; 8 months
  Incidence of adverse events as defined by REGULATION (EU) 2017/745(MDR) and MDCG 2020-10/1

CONTACTS AND LOCATIONS:
Overall Officials: Stefan De Wachter, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No